CLINICAL TRIAL: NCT02830035
Title: Comparison Between Real-Time Ultrasound Guidance vs Anatomical Landmark Technique on the Efficacy of Paramedian Spinal Anaesthesia
Brief Title: Real-Time Ultrasound-guidance Facilitates Paramedian Spinal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Soon Eu Chong, Medical Lecturer in Anesthesiology, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USM/JEPeM/283.2.(5)
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Wounds and Injuries
Keywords: ultrasound guided; spinal anesthesia; neuraxial block; paramedian
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anatomical Landmark Technique (Active Comparator): Traditional anatomical landmark technique based paramedian spinal anesthesia
  Interventions: Procedure: Anatomical Landmark Technique
- Real-time Ultrasound-guided Technique (Active Comparator): Ultrasound-guided paramedian spinal anesthesia Intervention: Ultrasound-guided Technique
  Interventions: Procedure: Real-time Ultrasound-guided

INTERVENTIONS:
Procedure: Real-time Ultrasound-guided — Real-time ultrasound guided paramedian spinal anesthesia
  Arms: Real-time Ultrasound-guided Technique
Procedure: Anatomical Landmark Technique — Conventional anatomical landmark technique for paramedian spinal anesthesia
  Arms: Anatomical Landmark Technique

SUMMARY:
The purpose of this study is to compare the clinical efficacy of real-time ultrasound guidance on spinal anesthesia vs the traditional anatomical landmark technique, by comparing success rate of spinal needle insertion, success rate rate of single needle pass, duration and immediate complications.

DETAILED DESCRIPTION:
Research hypothesis

1. Ultrasound guidance will lead to a significantly different success rate of paramedian spinal needle insertion, as well as the success rate of single-needle-pass when patient lying in lateral position.
2. Ultrasound guidance of paramedian spinal anaesthesia has a different rate of complication of spinal anaesthesia, e.g. postdural puncture headache and bloody taps.
3. Ultrasound guidance of paramedian spinal anaesthesia will cause a significant different in duration of giving spinal anaesthesia, compared to non ultrasound guided technique.

Justification of the Study

Ultrasound guidance in neuraxial blockade has been shown to be superior to palpation in correctly identifying lumbar intervertebral level, as well as improve efficiency and reduce complication of spinal anaesthesia.

Paramedian approach to the subarachnoid spaces is useful in situations where the patient's anatomy does not favor the midline approach, e.g., inability to flex the spine or heavily calcified interspinous ligaments. Studies have shown that choice of midline or paramedian approach did not affect the success rate of the subarachnoid puncture in general. Therefore, this is a technique that worth to be studied.

Orthopedic surgeries involving lower limbs are a common, in which many of the patients might be unable to sit up due to pain.

This study is mainly focused to access the optimal approach of doing paramedian approach of spinal anaesthesia in the condition when patient is lying lateral, in lower limb surgeries, as there is no local data that is available for our population. This will help to improve quality of anaesthesia in terms of patient satisfaction, as well as reduce complication.

Study setting: Operation theater, Hospital Universiti Sains Malaysia. Time frame: 12 months Population : Patients undergoing elective or emergency lower limb surgeries. On-site audit: Human Research Ethics Committee USM (HREC) Standard Operating Procedures will be according to guidelines of Human Research Ethics Committee USM (HREC)

Sample size determination

Sample size calculation was guided by Dr. Yee Cheng Kueh (Lecturer, Unit of Biostatistics and Research Methodology, School of Medical Sciences, Universiti Sains Malaysia) using Power and Sample size calculation software.

Sample size was based on previous literature by WANG et al comparing Real-time Ultrasound-assisted And Non-ultrasound-assisted Approach in combined spinal-epidural puncture obese patient. Sample size was calculated for primary outcome 1 (success rate of spinle needle insertion) and 2 (success rate of single needle pass), and secondary outcome 1 (duration for successful dural puncture and duration for procedure). The largest sample size was taken.

Methodology:

1. After approval from Human Research Ethics Committee USM (HREC), patient will be selected according to inclusion & exclusion criteria during preoperative assessment, from emergency or elective OT list.
2. Explain procedure to patient and get the written consent from patient.
3. Consented patients will be randomized into 2 arm: group U (ultrasound guided) and group P (anatomical landmark technique by palpation) using block randomization method and allocation concealment as:

   * 6 ballot cards will be put inside the envelope. Each of the cards state 6 different sequences of grouping (UUPP, PPUU, UPUP, PUPU, UPPU, and PUUP).
   * 1 card will be randomly taken each time by the nurse who assists anaesthesia to decide the group for the first four patients. This will be followed by other cards until all 6 sequences are completed. This means that at the end of 6 randomized sequences, there will be an equal 12 patients in each groups with the total number of 24 samples.
   * The randomization will be continued again as above until the total samples of collection are completed. (15x4 =60)
4. The monitoring of all patients will be standardized :

   * Noninvasive blood pressure (NIBP)
   * Heart Rate (HR)
   * Oxygen saturation , SPO2
   * Electrocardiogram (ECG)
5. Hemodynamic parameters such as systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), heart rate (HR) will be recorded before procedure, and post spinal 1min, 3 min, 5 min & 10 min.
6. Patient will then be positioned laterally with the operation limb on the dependent site.

   1. In the ultrasound group, a pre-procedural scan of the lumbar spine will be performed using portable ultrasound machine, Mindray M5 (Mindray, Shenzhen, China) with 2.5-3.0 MHz transducer.

      After aseptic skin preparation and draping, the convex 2.5-3.0MHz transducer will be covered with a sterile sheath. Sterile ultrasound gel will be used for transducer-skin contact.

      When the preferred lumbar interspace is in view on monitor, local anaesthetic (lignocaine 2% 2-3ml) will be infiltrated to the skin and underlying tissue 1-2 cm lateral to the identified spinous process. Under real-time ultrasound guidance, a spinal needle introducer is then inserted in-plane to the ultrasound probe, followed by A 25G Pencan® pencil point spinal needle.

      The backflow of cerebrospinal fluid (CSF) will confirmed a successful dural puncture.
   2. In the palpation group, the puncture site will be identified by palpation. The site where Tuffier's line (imaginary line between the iliac crests) crossed the spine is identified as level of L4 and the L3-4 or L4-L5 intervertebral space is chosen as the puncture site.

Once dural puncture is obtained, 2.5ml of isobaric bupivacaine and 25mcg of preservative-free fentanyl was injected.

Data will be analyzed using SPSS software.

For primary outcome 1 (success rate of spinle needle insertion), data obtained in the study will be analyzed with uncorrected chi-square test for comparison between Group Ultrasound and Group Palpation. Fisher's exact test was used in cases where assumption of Chi square was not met.

For primary outcome 2 (success rate of single needle pass), data obtained in the study will be analyzed with uncorrected chi-square test for comparison between Group Ultrasound and Group Palpation. Fisher's exact test was used in cases where assumption of Chi square was not met.

For secondary outcome 1 (duration for successful dural puncture and duration for procedure), data obtained will be analyzed with independent t-test for comparison of duration between Group Ultrasound and Group Palpation.

For secondary outcome 2 (immediate complication), data obtained will be analyzed descriptively as sample size will be too big to significantly compare the complication rates and was not cost effective.

ELIGIBILITY:
Inclusion Criteria:

* Consented adults aged at least 18 years old.
* ASA I to III.
* Presented for lower limb surgery.
* Fasted for at least 6 hours.

Exclusion Criteria:

* Patient refusal
* Contraindication to neuraxial block.
* Patient on anticoagulant medication, or coagulopathy (INR > 1.5)
* Patient on double antiplatelet, or thrombocytopenia (platelet < 100)
* Local infection at site of injection
* Indeterminate neurological disease
* Allergy to local anaesthetics
* Spinal abnormality
* Pregnancy.
* Previous surgery to lumbar region.
* BMI > 30

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
success rate of spinal needle insertion | during the procedure of spinal anesthesia
  The ability of getting a successful spinal anesthesia with a single skin puncture regardless of needle redirection.
success rate of single needle pass | during the procedure of spinal anesthesia
  The ability of getting a successful spinal anesthesia with a single skin puncture and no needle redirection.

SECONDARY OUTCOMES:
duration of procedure | during the procedure of spinal anesthesia
immediate complication | immediately after and within 1 week after given spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Soon Eu Chong, MD, MMed, Principal Investigator — Universiti Sains Malaysia; Mohd Nikman Ahmad, MD, MMed, Study Chair — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Niazi AU, Chin KJ, Jin R, Chan VW. Real-time ultrasound-guided spinal anesthesia using the SonixGPS ultrasound guidance system: a feasibility study. Acta Anaesthesiol Scand. 2014 Aug;58(7):875-81. doi: 10.1111/aas.12353. Epub 2014 Jun 18. PMID 24943307
- [Background] Ansari T, Yousef A, El Gamassy A, Fayez M. Ultrasound-guided spinal anaesthesia in obstetrics: is there an advantage over the landmark technique in patients with easily palpable spines? Int J Obstet Anesth. 2014 Aug;23(3):213-6. doi: 10.1016/j.ijoa.2014.03.001. Epub 2014 Mar 12. PMID 24768303
- [Background] Grau T, Leipold RW, Fatehi S, Martin E, Motsch J. Real-time ultrasonic observation of combined spinal-epidural anaesthesia. Eur J Anaesthesiol. 2004 Jan;21(1):25-31. doi: 10.1017/s026502150400105x. PMID 14768920
- [Background] Horlocker TT, Wedel DJ, Benzon H, Brown DL, Enneking FK, Heit JA, Mulroy MF, Rosenquist RW, Rowlingson J, Tryba M, Yuan CS. Regional anesthesia in the anticoagulated patient: defining the risks (the second ASRA Consensus Conference on Neuraxial Anesthesia and Anticoagulation). Reg Anesth Pain Med. 2003 May-Jun;28(3):172-97. doi: 10.1053/rapm.2003.50046. No abstract available. PMID 12772135
- [Background] Wang Q, Yin C, Wang TL. Ultrasound facilitates identification of combined spinal-epidural puncture in obese parturients. Chin Med J (Engl). 2012 Nov;125(21):3840-3. PMID 23106885
- [Background] Conroy PH, Luyet C, McCartney CJ, McHardy PG. Real-time ultrasound-guided spinal anaesthesia: a prospective observational study of a new approach. Anesthesiol Res Pract. 2013;2013:525818. doi: 10.1155/2013/525818. Epub 2013 Jan 10. PMID 23365568
- [Background] Brinkmann S, Tang R, Sawka A, Vaghadia H. Single-operator real-time ultrasound-guided spinal injection using SonixGPS: a case series. Can J Anaesth. 2013 Sep;60(9):896-901. doi: 10.1007/s12630-013-9984-9. Epub 2013 Jun 19. PMID 23780883
- [Background] Chin KJ, Perlas A, Chan V, Brown-Shreves D, Koshkin A, Vaishnav V. Ultrasound imaging facilitates spinal anesthesia in adults with difficult surface anatomic landmarks. Anesthesiology. 2011 Jul;115(1):94-101. doi: 10.1097/ALN.0b013e31821a8ad4. PMID 21572316